CLINICAL TRIAL: NCT04302090
Title: Changes in Pain Level With the Use of the Regulated Expiratory Method During Childbirth Process .
Brief Title: Changes in Pain Level With the Use of the Regulated Expiratory Method.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Kaouther Dimassi, associate professor obstetrics and gynecology faculty of medicine Tunis, University Tunis El Manar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Doloris-Winner-flow-URO-MG
Record Dates: First submitted 2020-03-05; First posted 2020-03-10 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Childbirth Process
Keywords: pain; childbirth; delivery; expiration; exercise; mothers
MeSH Terms: conditions — Pain; Death; Motor Activity

STUDY DESIGN:
Intervention Model Description: Each participant will experience successives periods A period of 4 consecutive contractions without using the expiration mouthpiece and a second period of 4 consecutive contractions using the the expiration mouthpiece .
  pain levels measured in each period will be compared for the same participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pain level changes according to the use of the Winner flow (Experimental): each included patient will experience :
  * a period of consecutive spontaneous uterine contractions without using the regulated expiration mouthpiece
  * a period of consecutive uterine contractions managed by the regulated expiration method using the Winner flow
  Interventions: Other: Regulated expiratory method

INTERVENTIONS:
Other: Regulated expiratory method — This method was originally a postpartum abdomino-perineal rehabilitation technique. It allows a functional abdominal rehabilitation by combining a regulated breath in a specific mouthpiece and an abdominal stimulation triggered by this same breath. The use of this method was extended to labor and childbirth. In fact, the application of the method during labor is based on the use of a flow regulating device (Winner Flow + URO-MG®). By regulating the flow of breath during a uterine contraction, it allows better pain management.
  Other Names: Winner flow Pro

SUMMARY:
Historically, pain management during childbirth has been a primary concern in the obstetric community. In recent decades, childbirth care providers have been witnessing, especially in developed countries, a real revolution in terms of approaches around this unique moment of birth. This is how perinatal professionals are no longer concerned only with medical follow-up and the smooth running of pregnancy or the well-being of the newborn, but also with overall support for women by promoting their active participation in the childbirth process. To this end, several methods of pain management are offered to women during labor. The more documented are: locoregional (epidural) anesthesia and acupuncture. These two methods are rarely available in Tunisian public maternity hospitals where 80% of deliveries are managed. In addition, Childbirth training workshops, psychoeducation and psychosocial couple-based programs are not available in tunisian public maternities. For example, only one public structure offers a painless delivery program at Farhat Hached Sousse hospital.

In consequence, women arriving at the labor room, are largely unaware of the basic principles of childbirth process. They do not know how to manage their pain.

the application of the GUILLARME® method during labor is based on the use of a flow regulating device (Winner Flow + URO-MG®). By regulating the flow of breath during a uterine contraction, it allows better pain management. Despite a positive feedback not only from parturients but also from midwives who practiced this method, actually investigators have only subjective evaluation with no real measurable and objective impact on pain levels during childbirth process. Consequently, investigators are conducting this scientific study whose main objective is:

-To evaluate changes in pain level with the use of regulated expiratory method during childbirth process.

DETAILED DESCRIPTION:
Historically, pain management during childbirth has been a primary concern in the obstetric community. In recent decades,childbirth care providers have been witnessing, especially in developed countries, a real revolution in terms of approaches around this unique moment of birth. This is how perinatal professionals are no longer concerned only with medical follow-up and the smooth running of pregnancy or the well-being of the newborn, but also with overall support for women by promoting their active participation in the childbirth process. To this end, several methods of pain management are offered to women during labor. The more documented are: locoregional (epidural) anesthesia and acupuncture. These two methods are rarely available in Tunisian public maternity hospitals where 80% of deliveries are managed. In addition, Childbirth training workshops, psychoeducation and psychosocial couple-based programs are not available in tunisian public maternities. For example, only one public structure offers a painless delivery program at Farhat Hached Sousse hospital.

In consequence, women arriving at the labor room, are largely unaware of the basic principles of childbirth process. They do not know how to manage their pain.

In order to overcome this situation, we introduced the GUILLARME® method to the obstetric care unit at Mongi Slim la Marsa hospital in January 2018. This method was originally a postpartum abdomino-perineal rehabilitation technique. It allows a functional abdominal rehabilitation by combining a regulated breath in a specific mouthpiece and an abdominal stimulation triggered by this same breath. The use of this method was extended to labor and childbirth. In fact, the application of the GUILLARME® method during labor is based on the use of a flow regulating device (Winner Flow + URO-MG®). By regulating the flow of breath during a uterine contraction, it allows better pain management. Despite a positive feedback not only from parturients but also from midwives who practiced this method, actually investigators have only subjective evaluation with no real measurable and objective impact on pain levels during childbirth process. Consequently, investigators are conducting this scientific study whose main objective is:

-To evaluate changes in pain level with the use of regulated expiratory method during childbirth process.

ELIGIBILITY:
Inclusion Criteria:

* women with a Gestational age of at least 30 weeks of amenorrhea
* women with a Normal fetal heart rate before inclusion.
* women having regular uterine contraction before inclusion .

Exclusion Criteria:

* Refusal of participation
* Women requiring epidural anesthesia
* Women in an advanced stage of labor with a cervical dilation upon admission over 3 cm
* A medical contraindication to vaginal delivery .
* Intra uterine fetal demise.
* Previous participation to childbirth training workshops
* Women without regular uterine contraction .
* Gestational term <30 weeks
* fetal heart rate abnormalities

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
analgesia nociception index | 60 minutes for each participant
  continuously measured by a monitor during the hole childbirth process. investigators will compare measured indexes during the two periods ( with intervention and without intervention.
  An index value close to 100 corresponds to a prominent parasympathetic tone (low stress level, analgesia) and a value close to 0 corresponds to a prominent sympathetic tone (high stress level, nociception). In parturients during labor or postoperative awake patients in the recovery room, a negative linear relationship between analgesia nociception index and pain scores is documented.

SECONDARY OUTCOMES:
Patient's pain management experience | up to 12 hours In deed , For each recruited patient this outcome will be measured in minutes between onset of labor and delivery
  a questionnair Patient's pain management experience according to the use or no use of the expiration mouthpiece during childbirth process .
  estimation of Patient's pain management experience according to the use or no use of the expiration mouthpiece during childbirth process .
  Patient's pain management experience according to the use or no use of the expiration mouthpiece during childbirth process .
  estimation of patient's pain management experience according to the use or no use of the expiration mouthpiece during childbirth process using a questionnair

CONTACTS AND LOCATIONS:
Overall Officials: kaouther dimassi, MD, Principal Investigator — university tunis el manar , faculty of medicine Tunis, TUNISIA
Locations (1):
- Mongi Slim University Hospital, La Marsa, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No